CLINICAL TRIAL: NCT00296972
Title: A Randomized, Multicenter, phaseIIIB, Two Arm Study Evaluating the Tolerability of Peginterferon Alfa-2a Plus Ribavirin in Patients With Chronic Hepatitis C Genotype 1 Infection co-Infected With Human Immunodeficiency Virus Receiving HAART Versus Not Receiving HAART
Brief Title: Tolerability of Peginterferon Plus Ribavirin for Chronic Hepatitis C and HIV for Patients Receiving Antiretroviral Medication vs Not Receiving Antiretroviral Medication
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: not funded
Sponsor: University Health Network, Toronto (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML 18562A
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2007-04

CONDITIONS: Chronic Hepatitis C; HIV Infections
Keywords: peg interferon; ribavirin; HAART; HIV; Chronic Hepatitis C; Treatment Experienced
MeSH Terms: conditions — Hepatitis C, Chronic; HIV Infections | interventions — Ribavirin

INTERVENTIONS:
Drug: peg interferon plus ribavirin

SUMMARY:
The main purpose of this study is to compare the safety, effectiveness and tolerability of using Pegasys with Copegus in people who have both the hepatitis C virus (HCV) genotype 1 and HIV who continue taking HAART (highly active antiretroviral therapy) to those who discontinue taking HAART.

Canadian guidelines recommend that both HIV and HCV should not be treated at the same time as the medications needed to treat these two diseases may interact and that which disease to treat first is dependent on the CD4 count. In this study, the CD4 count must be over 350 cells and one must be stable on HAART before starting the study medication Pegasys in combination with Copegus.

DETAILED DESCRIPTION:
Since the introduction of highly active antiretroviral therapies (HAART), liver disease secondary to HCV infection has become a leading cause of morbidity and mortality in HIV/HCV co-infection. The influence of HCV co-infection on the progression of HIV has been less clear and the results have been conflicting. Studies conducted in the pre-HAART era did not find that HIV/HCV co-infection influenced the progression of HIV-induced immunodeficiency or death. Of four large studies conducted after HAART was introduced, two suggested a faster progression of HIV disease in the presence of HCV co-infection and two found no influence of HCV co-infection on overall mortality or progression of HIV disease. HCV may also negatively influence HIV disease in indirect ways, such as making the discontinuation of antiretroviral treatment more frequent because of an increased risk of liver toxicity.The morbidity and mortality resulting from the rapid progression of HCV infection in HIV-co-infected patients, particularly given the advances in HIV treatment that have improved the life expectancy of HIV-infected patients, support treating HCV infection in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C genotype 1 infection·
* Detectable plasma HCV-RNA Roche>1000copies/ml, >600IU/ml
* Chronic liver disease consistent with CHC infection on a biopsy obtained within the past 24 months
* Patients with cirrhosis or incomplete cirrhosis must have an abdominal ultrasound, CT scan, or MRI scan without evidence of hepatocellular carcinoma and a serum AFP <100 ng/mL within 2 months of randomization
* Patients with CD4 cell count ³ 350 cells /µL
* Patients on stable highly active antiretroviral therapy (HAART) for at least 12 weeks prior to baseline with the exception of patients receiving didanosine
* HIV-1 RNA is < 5000 copies/mL

Exclusion Criteria:

* IFN, pegylated interferons, viramidine, levovirin, or ribavirin therapy at any previous time
* Patients with evidence of active hepatitis B infection. ( presence of HbsAg)
* History or evidence of decompensated liver disease and/or a Child-Pugh score > 5, bleeding from esophageal varices, hepatic malignancy
* abnormal bloodwork ie absolute neutrophil <1,Hbg <110, Platelets <70,creatinine <50

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-07; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To compare the safety and tolerability of PEG-IFN with ribavirin in HIV/HCV co-infected patients who continue HAART therapy compared to those who discontinue HAART therapy in the first 12 weeks

SECONDARY OUTCOMES:
To compare the sustained virological response.

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Cooper, MD, Study Director — The Ottawa Hospital, On; Marianne Harris, MD, Study Director — St. Paul's Hospital, Vancouver B.C; Marina Klein, MD, Study Director — Hopital Royal-Victoria/Institut Thoracique de Montreal,Que; Mark Poliquin, MD, Study Director — Clinique Médicale L'Actuel; Steve Shafran, MD, Study Director — University of Alberta Hospital, AB; Anita Rachlis, MD, Study Director — Sunnybrook & Women's College HSC, On; Chris Fraser, MD, Study Director — Victoria, BC; Val Montessori, MD, Study Director — St. Paul's Hospital, Vancouver B.C; Benoit Trottier, MD, Study Director — Clinique Medicale L'Actuel, Que; John Farley, MD, Study Director — Winnepeg, MB
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada